CLINICAL TRIAL: NCT06445153
Title: Digitalized Clinical Decision Support for the Prevention of Postoperative Delirium (POD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: BARMER (Other); Technische Universität Berlin (Other); Freie Universität Berlin (Other); Universitätsklinik der Ruhr-Universität Bochum (Unknown)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Digi-POD
Record Dates: First submitted 2024-05-23; First posted 2024-06-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Delirium
Keywords: Clinical decision support system, Delirium risk factors, recommendations, surgery
MeSH Terms: conditions — Emergence Delirium | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Digi-POD is a multicenter, prospective, longitudinal intervention study in a before-and-after design with quantitative process analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control phase (No Intervention): Control phase: in this phase, all study patients receive the standard therapy of the respective study center.
- Intervention phase (Experimental): In this phase, the intervention with Digi-POD is made available as Clinical Decision Support System. The intervention consists of providing patients, relatives and caregivers with Digi-POD decision support for the prevention of delirium and treatment decisions for delirium in accordance with the recommendations from the guidelines in addition to the standard therapy of the respective study center.
  Interventions: Other: Intervention with clinical decision support system

INTERVENTIONS:
Other: Intervention with clinical decision support system — To this phase, patient data is automated and systematically analyzed in order to derive decision support based on current evidence and make it available to Digi-POD users (patients, relatives, nursing staff, doctors, other healthcare professionals).
  Arms: Intervention phase

SUMMARY:
The project aims to improve patient safety, reduce barriers to the implementation of current guideline recommendations, reduce workload in clinics, increase efficiency in work processes and close gaps in care. Subprojects regarding delirium are implementes as well.

DETAILED DESCRIPTION:
Postoperative delirium (POD) is the most common post-operative complication in the 70+ age group, affecting approximately fifteen percent of elderly patients. POD is characterized by impaired attention, awareness, and cognitive function. Both patients and their families are severely affected by the effects of this condition. While symptoms of POD occur during hospitalization, they have a critical impact on post-hospitalization quality of life, dependency on long-term care, and life expectancy.

The overarching goal of the Digi-POD project consortium is to develop a digital decision support system that makes current evidence-based guideline recommendations for POD machine-readable and allows automated, real-time validation against clinical data.

Sub-projects such as a point prevalence analysis on the incidence of delirium on 2 days at the Charité and a staff survey conducted by Aktionsbündnis Patientensicherheit e.V. in all study centers accompany this study.

Further substudies initiated by Charité Universitätsmedizin Berlin:

Two substudies (one feasibility study and one acceptance study) will be conducted using the prototype of the Clinical Brain Protection (CBP) application in Digi-POD patients at Charité.

Interviews and a review of project documentation to analyze obstacles and solution strategies for implementing data security/information security will be organized by Fraunhofer Fokus. The results will be incorporated into the Data Security project report.

ELIGIBILITY:
Study patients:

Inclusion Criteria:

* Age ≥ 70 years
* Male and female patients
* Patients who are insured through statutory health insurance
* Patients capable of giving consent for inclusion: by the patient, preoperatively
* Patients under guardianship for inclusion: written declaration of consent by guardian
* Operation (elective)

Exclusion Criteria:

* Insufficient language skills
* Moribund patients

Study relatives

Inclusion Criteria:

* Age ≥ 18 years
* Male and female relatives
* Relatives capable of giving consent for inclusion

Exclusion Criteria:

* Insufficient language skills
* No consent for data entry

Substudy of the Charité - University Berlin:

Inclusion criteria:

- All inpatients ≥ 18 years of age who have undergone delirium screening with a validated delirium screening instrument

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Guideline adherence | Up to five days
  Guideline adherence: proportion of guideline recommendations fulfilled per patient in the first five postoperative days. The guideline adherence rate up to postoperative day 5 (or earlier if the patient has already been discharged) is calculated as a simple division: Number of recommendations fulfilled by number of all recommendations (N=6). A guideline adherence rate of at least 4 out of 6 points (67%) per patient is considered clinically sufficient.
Postperative delirium- free days | Up to five days
  Number of postoperative delirium- free days within 5 days postoperatively per patient.

SECONDARY OUTCOMES:
Causes of delirium | Up to seven days
  Causes of postoperative delirium- within 7 days postoperatively per patient.
Changes of Electroencephalography | Participants will be followed up until the end of the operation, an expected average of 60 minutes
  Signals are measured by Electroencephalography Monitor.
Blood pressure | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Blood pressure is measured in millimeters of mercury. Drop in blood pressure, Digi-POD cutoff RR systolic below 20% of baseline from start of surgery to discharge ICU.
Pulse | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Heart rate (or pulse rate) is the frequency of the heartbeat measured by the number of contractions of the heart per minute.
Heart rhythm | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Heart rhythm is measured by an electrocardiogram used to evaluate heart frequencies.
Heart rate | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Heart rate is measured by an electrocardiogram used to evaluate the heart. Heart rate drop Digi-POD cutoff below 50 bpm from start of surgery to discharge ICU.
Oxygen saturation | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Oxygen saturation is measured by pulse oximetry.
Amount of dexmedetomidine | Participants will be followed up until the end of intensive care unit stay, an expected average of 3 days.
  If dexmedetomidine is administered by the attending physician, the information from the patient's dexmedetomidine medication chart is recorded.
Therapeutic measures against postoperative delirium (POD) | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Multicomponent/multimodal preventive measures to avoid POD are recorded by a questionnaire.
Team meetings on postoperative delirium (POD) | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Multicomponent team meetings to discuss preventive measures to avoid POD will be recorded by a questionnaire.
Delirium incidence | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Delirium incidence is measured with validated delirium scores.
Delirium duration | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Delirium duration is measured in days.
Proportion of patients with adequate adherence | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Proportion of patients with adequate (at least 4 out of 6 points) adherence to guidelines.
Proportion of patients with good adherence | Up to 7 postoperative days
  Proportion of patients with good (at least 5 out of 6 points) adherence to guidelines
Number of POD-free days in patients who achieved less than 80% adherence to the guidelines. | Up to 7 postoperative days
  Number of POD-free days in patients who achieved less than 80% adherence to the guidelines.
Guideline adherence | Up to 7 postoperative days
  Percentage of guideline recommendations fulfilled per patient in the first 7 postoperative days.
Number of POD-free days within 7 days | Up to 7 postoperative days
  Number of POD-free days within 7 days is measured postoperatively per patient:in
Delirium incidence within 7 days | Up to 7 postoperative days
  Delirium incidence in patients who received delirium screening with validated delirium scores twice a day in at least two shifts (per-protocol analysis)
Anxiety | Up to 5 postoperative days
  Anxiety is measured by Faces Anxiety Scale
Pain | Up to 5 postoperative days
  Pain is measured with validated pain scores, scoring form 0 (no pain) to 10 (highest pain).
Depth of sedation | Up to 5 postoperative days
  Depth of sedation is measured with the Richmond Agitation-Sedation Scale (RASS)
Functional performance | Up to 5 postoperative days
  Functional performance is measured with the Glagow Coma Scale
Concomitant medication | Up to 5 postoperative days
  Concomitant medication is measured in dosis per day.
Complications | Up to 7 postoperative days
  Postoperative procedures/therapies and complications classified according to Clavien-Dindo
Infection status | Up to 7 postoperative days
  Infection status is measured by chart review
Charlson comorbidity index (CCI) | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  The total score in the CCI is derived by summing the assigned weights of all comorbid conditions presented by the client. Higher scores indicate a more severe condition and consequently, a worse prognosis.
Change in cognitive status I | Up to 6 months
  Cognitive status is measured with validated scores.
Change in cognitive status II | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Cognitive status is measured with the MOCA in patients with positive and negative MiniCog.
Change in care level for BARMER patients | Up to 6 months
  Care level is measured by chart review.
Change in utilization of inpatient care | Up to 6 months
Change in Patient-Reported Outcomes Measures (PROMs) | Up to 3 months
  Patient-Reported Outcome Measures are recorded by PROM instruments.
Change in Patient-Reported Experience Measures (PREMs) | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Patient-Reported Experience Measures are recorded by PREM instruments.
Change in the result from the detailed geriatric assessment and the frailty scoring | Up to 6 months
  Frailty is measured by a modified Fried score.
Length of hospital stay | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Length of hospital stay is measured in days.
Length of intensive care unit stay | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Length of intensive care unit stay is measured in days.
Discharge type | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Discharge type is taken from the medical record.
Length of stay in the recovery room | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Length of stay in the recovery room is measured in hours.
Duration of surgery | Participants will be followed up until the end of operation, an expected average of 2 hours
  Duration of surgery is measured in minutes.
Duration of anesthesia | Participants will be followed up until the end of operation, an expected average of 2 hours
  Duration of anesthesia is measured in minutes.
Recommended therapies | Up to 6 months
  Recommended therapies (physiotherapy, memory consultation, nutritional counseling) are measured by physical assessments.
Incidence of Post Intensive Care Syndrome (PICS) | Up to 3 months
  Incidence of Post Intensive Care Syndrome (PICS) is measured by a composite of psychological, cognitive and functional scores.
Social data/Paragraph 21 data | Up to 6 months
  Health economic data according to cost of patient care (The §21 dataset (diagnoses and operation-codes).
Social data | Up to 6 months
  Evaluation of social data (pseudonymised) only for patients with statutory BARMER insurance and only with the patient's written consent to the processing of social data.
All-cause "mortality" | Up to 6 months
  Mortality is measured inhospital and during ths FU phase.
Direct cost data | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Direct care costs during inpatient treatment from the perspective of SHI (statutory health insurance).
Follow-up costs | Up to 6 months
  e.g. for outpatient/inpatient treatment, medication, remedies/aids and long-term care) from the perspective of statutory health insurance (SHI) and statutory long-term care insurance (LTCI)
Utilization of benefits | Up to 6 months
  Utilization of benefits from (statutory health insurance) (SHI) and statutory long-term care insurance (GPV) (in particular need for long-term care, outpatient/inpatient treatment)
Personnel resources during the hospital stay | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Personnel resources are measured by commitment time
Investment costs | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Costs are calculated with project data.
Maintenance costs | Participants will be followed up until the end of hospital stay, an expected average of 7 days
  Costs are calculated with project data.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (4):
- Germany (4):
  - Institut für Anästhesiologie und Schmerztherapie-Herz- und Diabeteszentrum NRW- Universitätsklinik der Ruhr-Universität Bochum, Bad Oeynhausen, Bochum
  - Department of Anaesthesiolgy and Intensive Care Medicine CCM/CVK, Charite- University Berlin, Berlin
  - CARITAS Klinik Maria Heimsuchung, Berlin
  - Klinikum im Friedrichshain - Vivantes - Netzwerk für Gesundheit GmbH, Berlin

IPD SHARING:
Plan to Share IPD: No